CLINICAL TRIAL: NCT06137482
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Intravenously or Subcutaneously Administered REGN13335, a Platelet-Derived Growth Factor-B Antagonist, in Healthy Adult Participants
Brief Title: A Study to See How Safe and Tolerable Different Doses of REGN13335 Are When Administered Intravenously (IV) or Subcutaneously (SC) to Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R13335-HV-2289
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- IV Cohort 1 Low Dose (Experimental): Randomized as described in the protocol
  Interventions: Drug: REGN13335; Drug: Matching Placebo
- IV Cohort 2 Mid Dose (Experimental): Randomized as described in the protocol
  Interventions: Drug: REGN13335; Drug: Matching Placebo
- IV Cohort 3 High Dose (Experimental): Randomized as described in the protocol
  Interventions: Drug: REGN13335; Drug: Matching Placebo
- IV Cohort 4 Higher Dose (Experimental): Randomized as described in the protocol
  Interventions: Drug: REGN13335; Drug: Matching Placebo
- IV Cohort 5 Highest Dose (Experimental): Randomized as described in the protocol
  Interventions: Drug: REGN13335; Drug: Matching Placebo
- SC Cohort 1 Low Dose (Experimental): Randomized as described in the protocol
  Interventions: Drug: REGN13335; Drug: Matching Placebo
- SC Cohort 2 High Dose (Experimental): Randomized as described in the protocol
  Interventions: Drug: REGN13335; Drug: Matching Placebo
- IV or SC Optional Cohort (Experimental): ≤ Highest IV or SC Dose as described in the protocol Randomized as described in the protocol
  Interventions: Drug: REGN13335; Drug: Matching Placebo

INTERVENTIONS:
Drug: REGN13335 — Administered intravenous (IV) or subcutaneous (SC), sequential ascending single dose
Drug: Matching Placebo — Administered IV or SC, sequential ascending single dose

SUMMARY:
This study is researching an experimental drug called REGN13335. This is the first time that REGN13335 will be given to people. This study will enroll healthy adults.

The aim of the study is to see how safe and tolerable REGN13335 is in healthy volunteers.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is present in the blood of study participants at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Has a body mass index between 18 and 32 kg/m^2, inclusive, at the screening visit
2. Is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, laboratory safety tests, and electrocardiograms (ECGs) performed prior to administration of study drug (ie, screening and baseline visit)

Key Exclusion Criteria:

1. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric or neurological disease, as assessed by the investigator

NOTE: Other Protocol Defined Inclusion / Exclusion Criteria Apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAE's) through the end of the study (EOS) visit | Baseline to day 113
Severity of TEAE's through the EOS visit | Baseline to day 113

SECONDARY OUTCOMES:
Concentrations of functional REGN13335 in plasma through the EOS visit | Baseline to day 113
Incidence of anti-drug antibodies (ADA) to single doses of REGN13335 over time | Baseline to day 113
Titer of ADA to single doses of REGN13335 over time | Baseline to day 113

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- New Zealand Clinical Research, Christchurch, Canterbury, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/